CLINICAL TRIAL: NCT06031259
Title: An Open-Label Extension for Subjects in Studies HGT-HIT-046 and SHP609-302 Evaluating Long-Term Safety of Intrathecal Idursulfase-IT Administered in Conjunction With Intravenous Elaprase® in Subjects With Hunter Syndrome and Cognitive Impairment
Brief Title: Extension Study of Idursulfase-IT Along With Elaprase in Children and Adults With Hunter Syndrome and Cognitive Impairment
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-609-3001; 2023-504127-90-00 (EU CTIS Number: EU CTIS Number)
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Hunter Syndrome
Keywords: Drug Therapy
MeSH Terms: conditions — Mucopolysaccharidosis II | interventions — idursulfase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Idursulfase-IT (Experimental): Participants will receive idursulfase-IT once monthly and weekly IV infusions of elaprase at the dose used in previous studies (HGT-HIT-045/SHP609-302) via IDDD until benefit is no longer derived from the treatment, or treatment is no longer tolerable, or up to approximately 4.8 years.
  Interventions: Drug: Idursulfase-IT; Drug: Elaprase

INTERVENTIONS:
Drug: Idursulfase-IT — Idursulfase-IT intrathecally via IDDD.
Drug: Elaprase — Elaprase IV infusion.

SUMMARY:
The study is an extension of two previous studies (HGT-HIT-046 [NCT01506141] and SHP609-302 [NCT02412787]). Participants must have completed one of the previous studies. The main aim of this study is to collect more information about the safety of the treatments, idursulfase-IT and elaprase, in children and adults with Hunter syndrome and cognitive impairment. Participants will receive the same treatment as in the previous studies.

DETAILED DESCRIPTION:
The drug being tested in this study is called idursulfase. Idursulfase is being tested for long term safety in participants with Hunter syndrome and cognitive impairment.

The study will enroll up to approximately 8 patients. Participants will receive idursulfase-IT via intrathecal drug delivery device (IDDD) once monthly along with elaprase intravenous (IV) infusion, weekly.

This multi-center trial will be conducted in France and Canada. The overall time to participate in this study is approximately 4.8 years.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must have completed end of study assessments in studies HGT-HIT-046 [NCT01506141] or SHP609-302 [NCT02412787] and received a clinical benefit from idursulfase-IT in the opinion of the investigator.
2. The participant, or participant's legally designated representative, must have been informed of the nature of this open-label extension and must have voluntarily signed an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved informed consent form after all relevant aspects of the study have been explained and discussed. Written consent of the participant's legally designated representative (if applicable) and the participant's consent/assent, as relevant, must be obtained.
3. The participant has continued to receive elaprase on a regular basis in studies HGT-HIT-046 or SHP609-302.

Exclusion Criteria:

1. The participant has experienced, in the opinion of the investigator, a safety or medical issue that contraindicates treatment with idursulfase-IT, including, but not limited to, uncontrolled seizure disorder, bleeding disorder, and clinically relevant hypertension.
2. The participant has clinically relevant intracranial hypertension.
3. The participant is enrolled in another clinical study, other than studies HGT-HIT-046 or SHP609-302, that involves clinical investigations or use of any investigational product (drug or [intrathecal/spinal] device) within 30 days prior to study enrolment or at any time during the study.

Ages: 3 Years to 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) by Type and Severity | Up to approximately 4.8 years
  An adverse event (AE) means any untoward medical occurrence in a participant or participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. The severity of AEs will be determined per the investigator's assessment.
Number of Participants with AEs Related to Idursulfase-IT | Up to approximately 4.8 years
  An AE means any untoward medical occurrence in a participant or participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. Any adverse event related to idursulfase-IT will be reported in this outcome measure.
Number of Participants with AEs Related to the IDDD | Up to approximately 4.8 years
  An AE means any untoward medical occurrence in a participant or participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. Any adverse event related to the IDDD will be reported in this outcome measure.
Number of Participants with AEs Related to Device Surgical Procedure | Up to approximately 4.8 years
  An AE means any untoward medical occurrence in a participant or participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. Any adverse event related to device surgical procedure will be reported in this outcome measure.
Number of Participants with AEs Related to IT Administration Process | Up to approximately 4.8 years
  An AE means any untoward medical occurrence in a participant or participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. Any adverse event related to IT administration process will be reported in this outcome measure.
Number of Participants with AEs Related to IV Elaprase Infusion | Up to approximately 4.8 years
  An AE means any untoward medical occurrence in a participant or participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. Any adverse event related to IV elaprase infusion will be reported in this outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- Canada (3):
  - M.A.G.I.C. Clinic, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Hospital for Sick Children, Toronto, Ontario
- Hopital Femme Mere Enfant, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No
Takeda does not provide access to Individual Participant Data when a study is in a very limited (small) study population due to participant privacy concerns such as potential reidentification of study participants.

REFERENCES:
- See also: To obtain more information on the study, click here on this link — https://clinicaltrials.takeda.com/study-detail/5684362136074625?idFilter=%5B%22TAK-609-3001%22%5D